CLINICAL TRIAL: NCT02416336
Title: Evaluation of Intraoperative Usage of Sentinella in Detecting Sentinel Lymph Nodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oncovision Inc (Industry)
Collaborators: California Pacific Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLN-USA-1
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Melanoma; Head and Neck Cancer; Breast Cancer
Keywords: sentinel lymph node; lymphoscintigraphy; intraoperative gamma camera
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Breast Neoplasms

ARMS (1):
- Sentinella intraoperative use (Experimental): Standard of care intraoperative protocol
  1. Localize SLN with the Gamma Probe for In vivo count
  2. Optional (time permitting during surgical prep). Image same SLN with Sentinella (Pre-incision)
  3. Surgically remove/excise localized SLN
  4. Ex vivo count - excised SLN with Gamma Probe
  5. In vivo background/roaming count with Gamma Probe
  6. Repeat step 1-5, until no SLNs are found with the Gamma Probe (negative reading)
  Sentinella intraoperative imaging protocol
  1. Survey surgical field/Post-excision control with Sentinella for remaining SLNs
  2. If focal uptake seen in step 1, search for these occult SLNs with Gamma Probe and remove localized additional SLNs
  3. Record information on data sheet for each excised SLN with Gamma Probe and Sentinella
  Interventions: Device: Sentinella Intraoperative imaging protocol

INTERVENTIONS:
Device: Sentinella Intraoperative imaging protocol — There is a "holding" time of 15-20 minutes after the lymph node is removed during which the node is further dissected, examined and prepared for pathological analysis. This occurs before the procedure is completed in case the surgeon determines that further surgical exploration or tissue removal is required.
  In this study, the investigators will use this holding time to collect images of the sentinel lymph node area using the Sentinella camera for this study. Therefore, participation in this study will not increase the subject's overall procedure time. However, if the Sentinella camera detects something that the standard imaging techniques have missed, such as an additional sentinel node, the surgeon will do further exploration and tissue removal as needed.

SUMMARY:
The aim of this study is to investigate whether the Sentinella camera improves intraoperative detection and removal of sentinel lymph nodes (SLNs) when used in conjunction with standard detection methods. Of primary interest is whether the Sentinella camera identifies additional tumor-positive SLNs that are missed using traditional imaging techniques. Other outcomes related to the standard of care use of the Sentinella camera may also be assessed.

DETAILED DESCRIPTION:
Sentinella is an FDA-approved, high-resolution, portable gamma camera that gives valuable visual guidance to surgeons in certain types of cancer surgeries where no, or only limited, visual guidance was possible previously. The significance of this new aid is the improved possibility of locating and removing all lymph nodes that drain directly from tumors-so-called "SLNs"-in order to accurately assess both the staging of the cancer as well as the best possible operative and post-operative treatment. Sentinella can confirm that no significant lymph nodes are missed and document this "clean field" on the patient's permanent record.

Usually, there is more than one SLN. False-negative SLN biopsy results may impair patient outcome for several reasons: missed nodes might lead to recurrence that can be potentially difficult to treat on occasions, involved nodes may be a potential secondary source of distant metastases, and understaging affects decisions about systemic therapy and specific radiation therapy. Missing SLNs is one of the main factors which increase the false-negative rates.

Sentinel node biopsy is undoubtedly the standard of care for breast cancer and melanoma because of the vital information the histological status of these nodes gives. Correct identification of these SLNs is challenging because of limitations of current preoperative imaging and the lack of visualization in the OR:

* What appears to be a single node in a preoperative lymphoscintigraphy or SPECT can turn out to be 2 or more different nodes that are close together. This is due to relatively low spatial resolution of these technologies.
* Structures can be "hidden" by other structures such as the principle tumor/injection site, making identification difficult or impossible. In these cases, Sentinella will discover the structure upon removal of the principle tumor and aid the surgeon in its removal.
* Currently used gamma probes give only audible and non-recorded aid to surgeons and can easily miss structures when they are more than 2 cm deep in tissue.

Sentinella gives additional visual information to surgical teams that can improve patient outcomes. It does not replace, but rather compliments current standard procedures, and it offers precise documentation of each step of the procedure to be kept permanently on the patient's record.

1. After standard injection of radiotracer and imaging are performed preoperatively, Sentinella can be used in the OR to identify the position of the structures and mark the skin for surgeon's reference.
2. Before removal, Sentinella can be used to visualize and quantify the radioactivity of each structure. This information is stored for future reference.
3. Upon removal of each structure, Sentinella can be used to verify ex-vivo the activity of the structure removed.
4. After removal and verification of all the structures planned, Sentinella is used to confirm that no active structure is left in and to document the resulting "clean field"

The current standard of care for surgical SLN biopsy involves use of a gamma probe. In this study, the investigators will prospectively collect Sentinella images obtained during this standard of care procedure and compare and correlate the findings with other standard of care imaging studies, and treatment and outcome information.

ELIGIBILITY:
Inclusion Criteria:

* All melanoma patients, with a Breslow thickness >1mm, who are seen at CPMC for sentinel node biopsy will be eligible to participate in this study provided that they have given consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The percentage of patients for whom Sentinella detects additional tumor-positive SLNs. | 1 year
  Primary endpoint The percentage of patients for whom Sentinella detects additional tumor-positive SLNs.

SECONDARY OUTCOMES:
Mean percentage of SLNs detected using pre-operative lymphoscintigraphy and/or SPECT/CT | 1 Year
  The mean percentage of excised SLNs among the total number of SLNs detected using preoperative lymphoscintigraphy and/or single-photon emission computed tomography (SPECT)/CT. This is to evaluate the percentage of intraoperatively found SLNs, which are preoperatively visualized by lymphoscintigraphy and/or SPECT/CT.
Additional SLNs per patient found using Sentinella | 1 Year
  The proportion of patients who have additional SLNs found and the mean number of additional SLNs found per patient. This is to evaluate in how many patients additional SLNs are found with Sentinella after negative gamma probe screening. (Label these additional nodes as: post-excision control/same location, near-injection-site, deeply located/low-uptake SLNs, etc.).
Mean Sentinella imaging time | 1 Year
  Mean time required to complete intraoperative imaging with Sentinella. (After the surgery, the total image acquisition time for that patient can be found on Sentinella's database.)

CONTACTS AND LOCATIONS:
Locations (1):
- California Pacific Medical Center - Pacific Campus, San Francisco, California, United States

REFERENCES:
- [Background] Stoffels I, Poeppel T, Boy C, Mueller S, Wichmann F, Dissemond J, Schadendorf D, Rosenbaum-Krumme S, Klode J. Radio-guided surgery: advantages of a new portable gamma-camera (Sentinella) for intraoperative real time imaging and detection of sentinel lymph nodes in cutaneous malignancies. J Eur Acad Dermatol Venereol. 2012 Mar;26(3):308-13. doi: 10.1111/j.1468-3083.2011.04057.x. Epub 2011 Mar 23. PMID 21429042
- [Background] Vermeeren L, Valdes Olmos RA, Klop WM, Balm AJ, van den Brekel MW. A portable gamma-camera for intraoperative detection of sentinel nodes in the head and neck region. J Nucl Med. 2010 May;51(5):700-3. doi: 10.2967/jnumed.109.071407. Epub 2010 Apr 15. PMID 20395319
- [Background] Hellingman D, de Wit-van der Veen LJ, Klop WM, Olmos RA. Detecting near-the-injection-site sentinel nodes in head and neck melanomas with a high-resolution portable gamma camera. Clin Nucl Med. 2015 Jan;40(1):e11-6. doi: 10.1097/RLU.0000000000000370. PMID 24662667